CLINICAL TRIAL: NCT06485375
Title: Electromiographic Evaluation and Skeletal Parameters of Patients Requiring Orthodontic Treatment: a Prospective Cross-sectional Study
Brief Title: Electromiographic Evaluation and Skeletal Parameters of Patients Requiring Orthodontic Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Other Study IDs: 2024-EMGSKELETAL
Record Dates: First submitted 2024-05-21; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Skeletal Malocclusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients requiring orthopedic/orthodontic
  Interventions: Diagnostic Test: EMG

INTERVENTIONS:
Diagnostic Test: EMG — Disposable bipolar surface electrodes will be used. The patient's skin will be clean with cotton gauze soaked in alcohol before electrodes placement to reduce skin impedance. The operator will palpate the muscle belly while the patient clenches his teeth and will position surface electrodes in parallel to the muscular fibres. Doing so the position of the electrodes results as follows: Masseters electrodes will be fixed parallel to the exocanthion-gonion line and with the upper pole of the electrode under the tragus-labial commissural line. Temporalis electrodes will be positioned along the anterior margin of the muscle (corresponding to the frontoparietal suture). Suprahyoid muscles electrodes will be placed in the submental area nearly 1 cm posterior to the mental symphysis, paramedian to the midline and lightly diverging. A reference electrode will be applied to the forehead of the patient.

SUMMARY:
The relationship between form and function within the craniofacial complex has been investigated by several Authors. However, there is still controversy regarding the different electromyographic activation patterns of the elevator muscles of the jaw. One particularly contentious area of enquiry is whether it is facial morphology that determines the strength of muscle activation, or whether a strong musculature can influence skeletal growth processes.

In light of the aforementioned considerations, the objective of the current clinical observational study was to investigate the potential correlation between the electromyographic activity of selected masticatory muscles (masseter, anterior temporalis and suprahyoid) and the craniofacial morphology of subjects under examination, with a particular focus on elucidating the mechanical advantage derived from different sagittal relationships between the maxillae. The electromyographic evaluation is carried out before the beginning of the orthodontic treatment (T0).

DETAILED DESCRIPTION:
The relationship between form and function within the craniofacial complex has been investigated by several Authors. However, there is still controversy regarding the different electromyographic activation patterns of the elevator muscles of the jaw. One particularly contentious area of enquiry is whether it is facial morphology that determines the strength of muscle activation, or whether a strong musculature can influence skeletal growth processes.

In light of the aforementioned considerations, the objective of the current clinical observational study was to investigate the potential correlation between the electromyographic activity of selected masticatory muscles (masseter, anterior temporalis and suprahyoid) and the craniofacial morphology of subjects under examination, with a particular focus on elucidating the mechanical advantage derived from different sagittal relationships between the maxillae. The electromyographic evaluation is carried out before the beginning of the orthodontic treatment (T0).

Muscle activity is commonly recorded by means of surface electromyography (sEMG). However, sEMG data can be affected by various artifacts, resulting in questionable interpretation of the results. A standardisation procedure allows to reduce variability of the assessment of masticatory muscle activity during static and dynamic tasks.

Doing so the position of the electrodes results as follows:

* Masseters electrodes will be fixed parallel to the exocanthion-gonion line and with the upper pole of the electrode under the tragus-labial commissural line.
* Temporalis electrodes will be positioned along the anterior margin of the muscle (corresponding to the frontoparietal suture).
* Suprahyoid muscles electrodes will be placed in the submental area nearly 1 cm posterior to the mental symphysis, paramedian to the midline and lightly diverging.

A reference electrode will be applied on the forehead of the patient. The sEMG analysis will be composed of four parts:

1. Masticatory muscle standardisation procedures (repeated thrice): two 10 mm thick cotton rolls will be positioned on the mandibular posterior teeth of each participant, and a 5 second maximum voluntary contraction will be recorded to standardize anterior temporalis and superficial masseters sEMG signals. The mean sEMG potential obtained in the first acquisition was set at 100%, and all further ssEMG potentials will be expressed as a percentage of this value (μV/μV × 100).
2. Maximum voluntary teeth clenching: patients will be asked to clench their teeth in maximum intercuspation as hard as possible for 5 seconds.
3. Submental muscle standardisation procedures: participants will be asked to push their tongue against the palate (without teeth clenching), and a 5 seconds sEMG suprahyoid muscles activity will be recorded. All further sEMG potentials will be expressed as a percentage of this value (μV/μV × 100).
4. Saliva swallowing: participants will be asked to keep their mouth open to accumulate saliva and, when needed, to swallow "freely" (as usual) and a 5 seconds sEMG activity will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients needing an orthopaedic and/or orthodontic treatment
* Deciduous, mixed, or permanent dentition

Exclusion Criteria:

* Systemic diseases or congenital anomalies affecting craniofacial growth or development
* Signs or symptoms of temporomandibular disorder (TMD)
* Dental Pain
* Past maxillofacial surgery

Ages: 6 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients willing to begin orthopedic/orthodontic treatment
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-03 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-25 (Estimated)

PRIMARY OUTCOMES:
Percentage Overlapping Coefficient - POC % | Baseline (T0)
  It indicates in % the ratio between the activation of the left muscle compared to the right one and its value is between 0 and 100%. A POC of 100% identifies two muscles that activate symmetrically. A lower value shows a greater asymmetry of muscles activation. 95% of subjects without muscular imbalances of dental origin exhibits POC values between 80 and 90%. The POC detected are: Temporalis Anterioris, Masseter Muscle and mean.
Asymmetry index - ASIM % | Baseline (T0)
  It compares the influence of dental contacts on the total activity of the right MM and TA with respect to the left MM and TA. Its value varies between -100% and +100%. A negative value indicates a greater differential activity of the left muscles; conversely, a positive value indicates a greater differential activity of the right muscles. 95% of subjects without muscular imbalances of dental origin exhibits values of asymmetry between ± 10% .
Activation Index - ATTIV % | Baseline (T0)
  3.It compares the influence of dental contacts on the TA activity in relation to MM activity. A negative value implies greater differential recruitment of TA, while a positive value implies greater differential recruitment of the MM. 95% of subjects without muscular imbalances of dental origin exhibits activation values between ± 10%.
TORQUE % | Baseline (T0)
  Torque measures the differential activity of the right TA and left MM in relation to the antagonist torque. A prevalence of the right TA and left MM muscles, or right MM and left TA, may result in twisting forces on the jaw resulting in laterodeviation. This index ranges between -100% and +100%. -100% indicates the total prevalence of left TA and right MM, + 100% indicates the total prevalence of right TA and left MM. 95% of subjects without muscular imbalances of dental origin exhibits torque values between ±10%.
IMPACT % | Baseline (T0)
  It quantifies the total muscular activity performed during MVC relative to the standardization clenching on cotton rolls.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, MSc, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.